CLINICAL TRIAL: NCT05082298
Title: Pilot Test of a Stepped-Care Approach for Dental Fear at Private Dental Clinics
Brief Title: Dissemination of a Brief Dental Fear Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1UG3DE029453-01-1; 1UG3DE029453-01 (NIH)
Record Dates: First submitted 2021-09-17; First posted 2021-10-18 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dental Fear

STUDY DESIGN:
Intervention Model Description: Piloting dissemination and feasibility of a two-step dental fear treatment at private practices in a large metropolitan city.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dental Fear Intervention (Experimental): All participants will receive a brief 2-step treatment for dental fear (Dental FearLess app, In-Chair Treatment)
  Interventions: Behavioral: Dental FearLess app; Behavioral: In-Chair Treatment Protocol

INTERVENTIONS:
Behavioral: Dental FearLess app — Dental FearLess, is a self-administered psychoeducational intervention that will be accessed by participants via their personal smart device (In other words, this is an online application in which investigators present information about dental procedures. The user selects the procedure on which they would like information and then views a brief video on the selected procedure. It uses evidence-based tools to help participants manage their thoughts, feelings, and behavior related to dental fear to reduce fear during encounters with dental professionals.
Behavioral: In-Chair Treatment Protocol — This session is a 1-hour-in-person Cognitive Behavioral Therapy (CBT) dental fear session by study staff at the dental office. Participants will practice managing their thoughts, behaviors, and/or feelings when exposed to stimuli that they report still fearing. After each practice situation, the mental health provider and participant discuss the disconfirmatory evidence generated by the situation.

SUMMARY:
Despite the fact that several efficacious interventions for dental fear exist, it continues to be among the most common, and least addressed phobias among individuals. This reality is largely due to dissemination, or lack thereof. Research is needed on how to disseminate and implement such treatment in a way that recognizes the barriers to accessing and entering treatment for dental fear. Using a collaborative care approach, the investigators will pilot test, for feasibility and acceptability, a brief 2-step dental fear intervention. The first step will be an app intervention for moderate-to-severe dental that can be accessed by participants on a mobile device. The second step will consist of a one-hour face-to-face CBT intervention for participants delivered by a mental health professional at their dentist's office.

DETAILED DESCRIPTION:
Dental fear is among the most common individual phobias, and has devastating effects on oral and physical health, as well as emotional well-being. The behavioral avoidance associated with dental fear leads to neglect of prophylactic care, more dental emergencies, increased pain and suffering for individuals, and greater financial burdens, both for patients and society at large. Treatment remains inaccessible to the vast majority of fearful patients. Extremely efficacious brief evidence-based interventions for dental fear have not been administered outside of the specialty clinics in which they were developed. This is despite the ubiquitous nature of dental fear and its well-document impact on public health. Further, none of these existing treatment models can be easily incorporating into dental practices (due to issues of logistics, credentialed providers, time, financial costs, and disruptions of workflow).

Research is needed on how to disseminate and implement such treatment in a way that recognizes the barriers to accessing and entering treatment for dental fear. The investigators propose to pilot test, for feasibility and acceptability, Dental FearLess, a brief, free, self-directed, computerized intervention for moderate-to-severe dental fear that can be implemented in the waiting room of dental offices. Patients reporting moderate-to-severe dental fear after completing Dental FearLess will be offered a follow-up 1-hour session that covers the same content in person. Clearly, the challenge at present is not how to treat dental fear to reduce the financial and human suffering burden to public health, but how to disseminate and implement Evidence Based Interventions (EBIs) for dental fear in a way that recognizes the rewards and barriers in the U.S. healthcare system.

Stepped-care interventions have demonstrated efficacy for other behavioral and emotional problems. The investigators aim to test whether such interventions are feasible and acceptable, for both dentists and patients, for dental fear. If the pilot evaluation shows promise, it can be tested in larger studies and, if effective, be more widely implemented in the normal course of dental practice. This could improve uptake and, ultimately, patient outcomes compared with existing psychosocial interventions for dental fear.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe dental fear
* 18 years of age or older
* Fluent and literate in English
* Access to a device with which they will be piloting the intervention.

Exclusion Criteria:

* Does not have moderate to severe dental fear
* 17 years of age or younger
* Does not speak English
* Does not have access to a device with which they would be piloting the intervention

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Usability of the Dental FearLess App | Usability measures will be collected within 24 hours of app completion
  A measure based on the System Usability Scale will assess participant feelings about the app. Each item is scored on a 1 to 5 Likert scale, with 7 of the 21 items reversed coded. Possible scores will range from 21 to 105 with higher scores indicating more favorable assessments regarding usability of the app
Usability of the In-Chair Intervention | Usability measures will be collected within 24 hours of receipt of in-chair treatment
  A measure based on the System Usability Scale will assess participants feelings about the in-chair intervention. Each item is scored on a 1 to 5 Likert scale, with 3 of the 16 items reversed coded. Possible scores range from 16 to 80, with higher scores indicating more favorable assessments regarding the usability of the intervention

SECONDARY OUTCOMES:
Dental Practice Retention | Up to 6 months from enrollment
  Behavioral data on dental appointment attendance, treatment adherence following intervention
Overall Effectiveness of 2-Step Model | Up to 6 months from enrollment
  Change in dental fear assessed via several indicators (self reported absolute fear,experiences of anxiety disconfirmation, cognitions and affect experienced during next scheduled dental appointment)
Global Dental Fear | Assessed within the 24 hours before and within the 24 hours after app use.
  Gatchel's dental fear item will be used during screening for its brevity. Participants rate their dental anxiety/fear on a 0 (none) to 10 (high) scale.
Appointment Post-Survey | Assessed within 24 hours after using the app.
  Dental visit experience and fear-belief confirmation or disconfirmation questions.

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Heyman, PhD, Principal Investigator — New York University
Locations (2):
- United States (2):
  - Noble Dental Care, PC, Brooklyn, New York
  - Allen & Schwarz Dental, New York, New York

IPD SHARING:
Plan to Share IPD: No